CLINICAL TRIAL: NCT00012194
Title: Phase I Dose Escalation Study of UCN-01 (NSC 638850) Plus Cisplatin in Advanced Malignant Solid Tumors
Brief Title: 7-hydroxystaurosporine and Cisplatin in Treating Patients With Advanced Malignant Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03129; DMS 9934; DMS-9934; NCI-2331; NCT00227396 (obsolete NCT alias)
Record Dates: First submitted 2001-03-03; First posted 2003-01-27 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2013-07

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — 7-hydroxystaurosporine; Cisplatin

ARMS (1):
- Treatment (7-hydroxystaurosporine, cisplatin) (Experimental): Patients receive cisplatin IV over 1 hour on day 1 and UCN-01 IV continuously over 36-72 hours on day 2. Treatment repeats every 4 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: 7-hydroxystaurosporine; Drug: cisplatin; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: 7-hydroxystaurosporine — Given IV
  Other Names: UCN-01
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase I trial to study the effectiveness of combining UCN-01 with cisplatin in treating patients who have advanced solid tumors. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. UCN-01 may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth and may help cisplatin kill more cancer cells by making tumor cells more sensitive to the drug.

DETAILED DESCRIPTION:
OBJECTIVES:

I. To establish the maximum tolerated dose (MTD) of cisplatin in combination with UCN-01 in patients with advanced malignancies.

II. To assess the toxicity and observe the potential antitumor activity of UCN-01 plus cisplatin in advanced malignancies at each dose level studies.

III. To determine the pharmacokinetics of UCN-01 and cisplatin on this treatment schedule.

IV. To perform laboratory correlative studies to investigate intermediate molecular markers of the activity of UCN-01 and cisplatin at the cellular level.

OUTLINE: This is a dose-escalation study of cisplatin.

Patients receive cisplatin IV over 1 hour on day 1 and UCN-01 IV continuously over 36-72 hours on day 2. Treatment repeats every 4 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of cisplatin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed every 2-3 months for at least 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Advanced or metastatic, histologcally/cytologically confirmed malignant solid tumor, not expected to clinically benefit from standard therapy
* Life expectancy greater than 3 months
* Previous chemotherapy and/or radiotherapy must have been completed at least four weeks (six weeks for prior treatment with mitomycin or nitrosoureas) and patients should have recovered from all toxicities of that therapy before treatment under this protocol
* All patients must have recovered from any surgical procedure
* Serum creatinine must be within the institutional limits of normal and an estimated creatinine clearance of >= 60 ml/min
* Normal bilirubin is required
* SGOT/AST must be less than or equal to 2.5 times the upper limit of institutional normal
* WBC >= 4000/mm^3
* Absolute neutrophil count >= 2000/mm^3
* Platelet count >= 150,000/mm^3
* Patients must have a Karnofsky Performance Status of 60% or greater
* Subjects who are fertile must use a medically acceptable contraceptive throughout the treatment period and for three months following cessation of treatment; subjects must be made aware, before entering this trial, of the risk in becoming pregnant or in fathering children
* A signed informed consent (approved by the IRB) must be obtained prior to trial entry
* Tumor site accessible for both pre-treatment and post-treatment biopsy is preferred during dose-finding, and is required for patients entering the expanded cohort at the MTD
* All patients require a central indwelling venous catheter prior to treatment under this protocol

Exclusion Criteria:

* Peripheral neuropathy > grade I
* Any prior mediastinal radiotherapy
* Any history of coronary artery disease
* Class III or IV congestive heart failure according to the New York Heart Classification
* History of allergic reactions to appropriate diuretics or antiemetics (e.g., 5-HT3 antagonists) to be administered in conjunction with protocol directed chemotherapy
* Brain metastasis
* Uncontrolled intercurrent illness that would preclude tolerance and completion of the protocol treatment, including vigorous hydration prior and subsequent to cisplatin therapy
* Lactating or pregnant women are excluded to avoid potential harm to the unborn child or infant; documentation of a negative, serum beta-HCG pregnancy test must be available for pre-menopausal women with intact reproductive organs and for women less than two years after menopause
* Receipt of any investigational drug within 30 days before beginning treatment with study drug
* Medical, social, or psychological factors that would prevent the patient from completing the treatment protocol
* Patients with clinically significant hearing loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2001-03; Primary Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
MTD of cisplatin defined as the highest dose level in which six patients have been evaluated for toxicity with no more than one patient experiencing DLT attributable to the study drugs | 4 weeks
  Graded using the NCI CTCAE.
Toxicity observed at each dose level, graded using the NCI CTCAE | Up to 7 years
  Summarized in terms of type, severity, time of onset, duration, and reversibility or outcome.

SECONDARY OUTCOMES:
Objective tumor response | Up to 7 years
  Summarized at each dose level, and the number and percent responding combined across dose levels.
Overall survival | From registration to time of death due to any cause, assessed up to 7 years
  Summarized with Kaplan-Meier plots.
Time to treatment failure | From registration to the first observation of disease progression, death due to any cause, or early discontinuation of treatment, assessed up to 7 years
  Summarized with Kaplan-Meier plots.
Duration of response | Up to 7 years
  Summarized with Kaplan-Meier plots.

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Perez, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States